CLINICAL TRIAL: NCT02379728
Title: A Maternal Device to Reduce the Risk of Stillbirth and Low Birth-Weight
Brief Title: Ghana PrenaBelt Trial: A Positional Therapy Device to Reduce Still-Birth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Allan Kember (Other)
Collaborators: Korle-Bu Teaching Hospital, Accra, Ghana (Other); Grand Challenges Canada (Other); Innovative Canadians for Change (Other); Global Innovations for Reproductive Health and Life (Other); Kaishin Chu Design (Industry)
Responsible Party: Sponsor-Investigator, Allan Kember, Medical Student, IWK Health Centre
Organization: IWK Health Centre (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: GCC-S7-0629-01-10-ACC; FDA/CT/152 (Other: Ghana Food and Drugs Authority)
Record Dates: First submitted 2015-02-18; First posted 2015-03-05 (Estimated); Results first posted 2020-04-02 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Sleep; Pregnancy; Stillbirth; Infant, Low Birth Weight; Infant, Small for Gestational Age; Infant, Very Low Birth Weight; Fetal Growth Retardation; Fetal Hypoxia
Keywords: positional therapy; tennis ball technique; sleep pregnancy; supine position; supine; sleep position; low birth weight; stillbirth; intrauterine growth restriction
MeSH Terms: conditions — Stillbirth; Fetal Growth Retardation; Fetal Hypoxia; Deception

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- PrenaBelt (Experimental): Participants will be instructed to use the PrenaBelt nightly for the remainder of their pregnancy in addition to receiving the local standard of care.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
  Interventions: Device: PrenaBelt
- PrenaBelt with Body Position Sensor (Experimental): Participants will be instructed to use the PrenaBelt (with integrated body position sensor (BPS)) nightly for the remainder of their pregnancy in addition to receiving the local standard of care. The BPS will be securely integrated into a small pocket on the PrenaBelt. The BPS is not expected to affect body position or sleep.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
  Interventions: Device: PrenaBelt; Device: Body Position Sensor
- Control (Sham Comparator): Participants will be instructed to use the sham-PrenaBelt nightly for the remainder of their pregnancy in addition to receiving the local standard of care.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
  Interventions: Device: sham-PrenaBelt
- Control with Body Position Sensor (BPS) (Sham Comparator): Participants will be instructed to use the sham-PrenaBelt (with integrated BPS) nightly for the remainder of their pregnancy in addition to receiving the local standard of care. The BPS will be securely integrated into a small pocket on the sham-PrenaBelt. The BPS is not expected to affect body position or sleep.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
  Interventions: Device: Body Position Sensor; Device: sham-PrenaBelt

INTERVENTIONS:
Device: PrenaBelt — The PrenaBelt (PB) is a belt-like, positional therapy (PT) device designed for pregnant women. While the PB does not prevent the user from lying on her back during sleep, it is expected to significantly decrease the amount of time a user spends supine via the mechanism of PT. PT is a simple, non-invasive, inexpensive, long-established, safe, and effective intervention for preventing people with positional-dependent snoring or obstructive sleep apnea from sleeping on their back - a position that exacerbates their condition.
  The PB is worn at the level of the waist or thorax. By design, the PB affects subtle pressure points on the user's back while supine, activating her body's natural mechanism to reposition itself to relieve discomfort, thereby reducing the amount of time spent supine.
  Arms: PrenaBelt; PrenaBelt with Body Position Sensor
Device: Body Position Sensor — The Body Position Sensor (BPS) is for research purposes only. The BPS can be securely integrated into a pocket on the PrenaBelt (PrenaBelt with BPS Arm) or sham-PrenaBelt (Control with BPS Arm). The BPS is a small, electronic data acquisition device. The BPS uses a three axes accelerometer to detect orientation of the PrenaBelt, and thus the user (right, left, prone, supine), in three-dimensional space. The accelerometer data is collected continually with time stamping and stored on the BPS hard drive and can be accessed via connecting it to a computer. The BPS is not expected to affect the body position of the user.
  Arms: Control with Body Position Sensor (BPS); PrenaBelt with Body Position Sensor
Device: sham-PrenaBelt — The PrenaBelt can be easily converted into a sham-PrenaBelt for research purposes by removing the hard balls from its pockets or exchanging these hard balls for soft balls so it cannot provide pressure points, i.e., positional therapy function. The sham-PrenaBelt looks, fits, and feels like the PrenaBelt but cannot provide positional therapy.
  Arms: Control; Control with Body Position Sensor (BPS)

SUMMARY:
Every day in Ghana, 47 babies are stillborn (SB) and 232 babies are born with low birth-weight (LBW) - many of whom will die in infancy or suffer lifelong consequences.

Sleeping on the back during pregnancy has recently emerged in scientific literature as a potential risk factor for SB and LBW. In fact, one of the earliest studies to demonstrate this link was conducted in Ghana by investigators on this protocol.

When a woman in mid-to-late-pregnancy lies on her back, her large uterus compresses one of the major veins that delivers blood back to her heart and may completely obstruct it. This may result in less blood being returned to her heart and less blood being pumped to her developing fetus. Such changes may negatively impact the growth of her fetus and, along with some other risk factors, may contribute to the death of her baby.

The investigators have developed a device, 'PrenaBelt', to significantly reduce the amount of time a pregnant woman spends sleeping on her back. The PrenaBelt functions via a simple, safe, effective, and well-established modality called positional therapy.

The purpose of this study is to determine the effect of the PrenaBelt on birth-weight and assess the feasibility of introducing it to Ghanaian third-trimester pregnant women in their home setting via an antenatal care clinic and local health-care staff. Data from this study will be used in effect size calculations for the design of a large-scale, epidemiological study targeted at reducing LBW and SB in Ghana and globally.

DETAILED DESCRIPTION:
Introduction:

According to the World Health Organization (WHO), stillbirth (SB) is defined as fetal death at gestation ≥28 weeks or weight ≥1000g. In addition to the loss of life for the stillborn baby, parents whose baby is stillborn must cope with the psychological grief of losing their baby, which results in markedly increased mortality in bereaved parents when compared with non-bereaved parents.

Low birth-weight (LBW) is defined as a weight less than 2500g at birth. LBW is a significant contributor to SB, and infants with LBW are 20 times more likely to die in the first year than heavier babies. Although LBW babies constitute only about 15% of live births, they account for 60-80% of neonatal deaths. Neonatal deaths (death within the first year of life) account for 40% of all deaths under the age of five years. LBW also accounts for significant morbidity such as cognitive impairment, and chronic diseases later in life. LBW arises through short gestation (preterm birth) or in-utero growth restriction, or both.

Women in Ghana suffer from one of the highest perinatal mortality rates in the world. Every day in Ghana, 47 babies are stillborn and 232 babies are born with LBW - many of whom will die in infancy or suffer lifelong consequences. As such, Ghana urgently requires inexpensive interventions to reduce perinatal morbidity and mortality - assisting pregnant Ghanaian women to avoid sleeping on their back might be one such intervention.

Background - Maternal Position:

In obstetrics, it is well-known that when a pregnant woman assumes the supine position (laying on her back) during the day, maternal cardiovascular parameters and/or fetal oxygenation are altered, occasionally causing significant fetal heart rate changes, particularly during labor. However, until recently, there has been little evidence on the effect of supine position during sleep in pregnancy. Recently, three studies have suggested that maternal sleep position may be a risk factor for SB and LBW. This is significant given that the majority of third trimester pregnant women spend up to 25% of their sleep time supine. In the Auckland Stillbirth Study, the population attributable risk (PAR) for non-left sleep position to SB was found to be 37%, which is greater than the PARs of the three most important modifiable risk factors for SB (obesity, advanced maternal age, and smoking) combined. In an African population, investigators on this protocol found that supine sleep during pregnancy was an independent predictor of LBW (OR, 5.0; 95% confidence interval (CI), 1.2-20.2; P=0.025) and SB (OR, 8.0; 95% CI, 1.5-43.2; P=0.016), when controlling for covariates maternal age, gestational age, parity, and the presence of pre-eclampsia. Notably, LBW was found to mediate the relationship between supine sleep and SB. Currently, there is much interest and follow up research occurring worldwide, with a growing body of evidence regarding the detrimental effects of supine sleep position on pregnancy outcomes.

One proposed model is that the maternal supine position during sleep is a stressor that plays a causative role in LBW and SB via compression of the abdominal aorta and inferior vena cava ('aortocaval compression'), resulting in negative sequelae. The investigators hypothesize that by mitigating this stressor, they may protect the fetus from LBW or SB.

Background - Maternal Device:

Given the emerging data suggesting that supine sleep may play a role in LBW and SB and the high perinatal mortality rate in Ghana, a simple intervention may allow the investigators to improve fetal outcomes.

Some pregnant women sleep with many pillows supporting their body, including a pillow behind their back to avoid the supine position. Asking women to sleep on their left increases the percentage of left sided sleep to approximately 60% of the night; however, this may come at a cost of a slightly reduced sleep duration, perhaps due to women feeling they need to make a conscious effort to maintain a certain sleep position.

Hence, a simple, low-cost, and easily-implemented device has been developed for use by pregnant women to mitigate this risk factor. The investigators anticipate that using this device will remove the need for the woman to make a conscious effort to avoid the supine sleeping position. The device name is 'PrenaBelt'. The PrenaBelt is currently at the prototype stage of development, and as such, this proposal is a proof-of-concept/feasibility project.

The PrenaBelt is a belt-like, positional therapy device designed specifically for pregnant women. While the PrenaBelt does not prevent the user from lying on her back during sleep, it is expected to significantly decrease the amount of time she spends in this position via the mechanism of positional therapy. Positional therapy is a simple, non-invasive, inexpensive, long-established, safe, and effective intervention for preventing people with positional-dependent snoring or mild to moderate obstructive sleep apnea from sleeping on their back - a position that exacerbates their condition.

The PrenaBelt is worn at the level of the waist. By virtue of its design and position on the user's body, the PrenaBelt affects subtle pressure points on the back of the user when she lies on her back. These subtle pressure points activate her body's natural mechanism to spontaneously reposition itself to relieve discomfort, thereby reducing the amount of time she remains on her back during sleep. The PrenaBelt is also designed for adjustability and comfort.

The investigators have designed an electronic Body Position Sensor (BPS) that can be securely integrated into a pocket on the PrenaBelt. The BPS will record body position of the user (left, right, prone, supine). The BPS is for research purposes only.

Study Design:

The feasibility (technical, operational, cultural), efficacy, acceptability, and compliance of the PrenaBelt intervention in the target population during the third trimester of pregnancy in an antenatal care clinic and home settings and the effect of PrenaBelt treatment on birth weight will be evaluated via a sham-controlled, double-blind, randomized controlled trial. Preliminary data will be collected for the design of a future, large-scale, parallel-group, randomized controlled trial to determine the efficacy of the PrenaBelt intervention in improving pregnancy outcomes in a resource-limited setting.

A small cohort of participants from the treatment and control groups will be randomly selected to use BPS's throughout the third trimester of pregnancy. Each BPS participant in the treatment group will be matched to a BPS participant in the control group using BMI (normal, overweight, obese) and age (within 5 years; 2.5 years each side) as matching variables and BPS data will be compared. These data will serve as preliminary objective evidence of PrenaBelt usage and effect on maternal sleeping position during the third trimester of pregnancy in the target population and setting.

Potential Harms:

This study is minimal risk. Participants in this study are at no greater risk of harms when completing the activities of this study than those risks they encounter in their everyday life.

The PrenaBelt, sham-PrenaBelt, and Body Position Sensor devices are non-invasive medical devices of Health Canada Class I designation. Pregnant women typically sleep with many pillows supporting their body, including a pillow behind their back to avoid the supine position. The PrenaBelt is a positional therapy device that may assist pregnant women to avoid supine sleep. Positional therapy devices have been shown to be safe and approved for use by humans by the US Food and Drug Administration. In addition, maternal body pillows, regular pillows, and pelvic belts (lumbar support) have been used by pregnant women during sleep without reports of serious adverse effects for the mother or neonate [Victoria Pennick and Sarah D Liddle, "Interventions for preventing and treating pelvic and back pain in pregnancy (Review)," The Cochrane Collaboration, London, Review 2013].

Participants in both the intervention and control groups may experience discomfort while learning to sleep with the PrenaBelt/sham-PrenaBelt, which theoretically may lead to delayed onset of sleep, arousals from sleep, and loss of sleep. Participants will be instructed how to, and told that they can, remove the PrenaBelt/sham-PrenaBelt and discontinue use at any time without penalty if they become too uncomfortable.

ELIGIBILITY:
Inclusion Criteria:

* ≥18 years old
* low-risk singleton pregnancy
* entering the last trimester of pregnancy (in range 26-30 weeks of gestation)
* residing in the Greater Accra Metropolitan Area or area served by the Korle Bu Teaching Hospital
* fluent in either English, Twi, or Ga.

Exclusion Criteria:

* BMI ≥ 35 at booking (first antenatal appointment for current pregnancy)
* pregnancy complicated by obstetric complications (hypertension [pre-eclampsia, gestational hypertension, chronic hypertension], diabetes [gestational or not], or intra-uterine growth restriction [<10th %ile for growth])
* sleep complicated by medical conditions (known to get <4 hours of sleep per night due to insomnia, or musculoskeletal disorder that prevents sleeping on a certain side [e.g., arthritic shoulder])
* multiple pregnancy
* known fetal abnormality
* maternal age >35

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 200 (Actual)
Dates: Start 2015-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Heather M Scott, MD FRCSC, Study Chair — The IWK Health Centre; Jerry Coleman, MB ChB FWACS, Principal Investigator — Korle Bu Teaching Hospital
Locations (1):
- Korle Bu Teaching Hospital, Accra, Greater Accra Region, Ghana

REFERENCES:
- [Background] Owusu JT, Anderson FJ, Coleman J, Oppong S, Seffah JD, Aikins A, O'Brien LM. Association of maternal sleep practices with pre-eclampsia, low birth weight, and stillbirth among Ghanaian women. Int J Gynaecol Obstet. 2013 Jun;121(3):261-5. doi: 10.1016/j.ijgo.2013.01.013. Epub 2013 Mar 15. PMID 23507553
- [Background] Stacey T, Thompson JM, Mitchell EA, Ekeroma AJ, Zuccollo JM, McCowan LM. Association between maternal sleep practices and risk of late stillbirth: a case-control study. BMJ. 2011 Jun 14;342:d3403. doi: 10.1136/bmj.d3403. PMID 21673002
- [Background] Gordon A, Raynes-Greenow C, Bond D, Morris J, Rawlinson W, Jeffery H. Sleep position, fetal growth restriction, and late-pregnancy stillbirth: the Sydney stillbirth study. Obstet Gynecol. 2015 Feb;125(2):347-355. doi: 10.1097/AOG.0000000000000627. PMID 25568999
- [Background] Platts J, Mitchell EA, Stacey T, Martin BL, Roberts D, McCowan L, Heazell AE. The Midland and North of England Stillbirth Study (MiNESS). BMC Pregnancy Childbirth. 2014 May 21;14:171. doi: 10.1186/1471-2393-14-171. PMID 24885461
- [Background] Warland J, Mitchell EA. A triple risk model for unexplained late stillbirth. BMC Pregnancy Childbirth. 2014 Apr 14;14:142. doi: 10.1186/1471-2393-14-142. PMID 24731396
- [Background] O'Brien LM, Warland J. Typical sleep positions in pregnant women. Early Hum Dev. 2014 Jun;90(6):315-7. doi: 10.1016/j.earlhumdev.2014.03.001. Epub 2014 Mar 21. PMID 24661447
- [Derived] Coleman J, Grewal S, Warland J, Hobson S, Liu K, Kember A. Maternal positional therapy for fetal growth and customised birth weight centile benefit in a Bayesian reanalysis of a double-blind, sham-controlled, randomised clinical trial. BMJ Open. 2024 Apr 28;14(4):e078315. doi: 10.1136/bmjopen-2023-078315. PMID 38684260
- [Derived] Coleman J, Okere M, Seffah J, Kember A, O'Brien LM, Borazjani A, Butler M, Wells J, MacRitchie S, Isaac A, Chu K, Scott H. The Ghana PrenaBelt trial: a double-blind, sham-controlled, randomised clinical trial to evaluate the effect of maternal positional therapy during third-trimester sleep on birth weight. BMJ Open. 2019 May 1;9(4):e022981. doi: 10.1136/bmjopen-2018-022981. PMID 31048420
- See also: Allan Kember's (Project Lead, Project Principal Investigator) blog - Project Updates — https://gojamverandah.wordpress.com/
- See also: Grand Challenges Canada - News Release — http://bit.ly/1ze8A0Z
- See also: Global Innovations for Reproductive Health and Life - Project Page — http://www.girhl.org/maternal-health-initiative/

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were recruited by maternity personnel when presenting for antenatal care at the Korle Bu Teaching Hospital. Between September 2015 and March 2016, 276 women were assessed for eligibility. Seventy-six (28%) did not meet the eligibility criteria. When the target enrollment (N=200) was reached, recruitment was stopped.
Groups:
- Control: Participants will be instructed to use the sham-PrenaBelt nightly for the remainder of their pregnancy in addition to receiving the local standard of care.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
  sham-PrenaBelt: The PrenaBelt can be easily converted into a sham-PrenaBelt for research purposes by removing the hard balls from its pockets or exchanging these hard balls for soft balls so it cannot provide pressure points, i.e., positional therapy function. The sham-PrenaBelt looks, fits, and feels like the PrenaBelt but cannot provide positional therapy.
Period: Overall Study
Arm/Group | PrenaBelt | PrenaBelt With Body Position Sensor | Control | Control With Body Position Sensor (BPS)
Started | 84 | 16 | 84 | 16
Completed | 78 | 16 | 74 | 13
Not Completed | 6 | 0 | 10 | 3
Not completed — Lost to Follow-up | 1 | 0 | 3 | 0
Not completed — Withdrawal by Subject | 5 | 0 | 5 | 3
Not completed — Protocol Violation | 0 | 0 | 2 | 0

BASELINE CHARACTERISTICS:
Population: 12 PrenaBelt and 7 sham participants excluded from analysis population. Two arms: PrenaBelt (participants with and without BPS) and Control (participants with and without BPS). BPS was not expected to affect body position. We did not intend readers would interpret this as 4 different treatments. No arms are missing from the entered data.
Groups:
- PrenaBelt: Participants will be instructed to use the PrenaBelt nightly for the remainder of their pregnancy in addition to receiving the local standard of care.
  A small subset of this group (n=16) will have a body position sensor (BPS) securely integrated into a small pocket on the PrenaBelt. The BPS is not expected to affect body position or sleep.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
- Control: Participants will be instructed to use the sham-PrenaBelt nightly for the remainder of their pregnancy in addition to receiving the local standard of care.
  A small subset of this group (n=16) will have a body position sensor (BPS) securely integrated into a small pocket on the sham-PrenaBelt. The BPS is not expected to affect body position or sleep.
  Participants will be followed by study personnel through the remainder of pregnancy and delivery.
- Total: Total of all reporting groups
Arm/Group | PrenaBelt | Control | Total
Number analyzed (Participants) | 82 | 80 | 162
Age, Continuous [Median (Inter-Quartile Range); unit: years] | 29 [27 to 31] | 29 [27 to 32] | 29 [27 to 32]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 82 | 80 | 162
  Male | 0 | 0 | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  Ghana | 82 | 80 | 162
Gestational age (weeks) [Median (Inter-Quartile Range); unit: weeks] | 28 [26.5 to 28.3] | 28 [27 to 29] | 28 [27 to 29]
Gravidity [Count of Participants; unit: Participants]
  Gravida 1 | 20 | 31 | 51
  Gravida ≥2 | 62 | 49 | 111
Parity [Count of Participants; unit: Participants]
  Para 0 | 29 | 38 | 67
  Para ≥1 | 53 | 42 | 95
Education [Count of Participants; unit: Participants]
  Tertiary | 50 | 48 | 98
  Vocational | 1 | 1 | 2
  Senior High | 15 | 26 | 41
  Junior High or less | 16 | 5 | 21
Household Income [Median (Inter-Quartile Range); unit: Cedis per month] — Average currency exchange rate for recruitment period: 1 United States Dollar (USD) = 3.84 Cedis Population: Some participants did not wish to disclose this information.
  Cedis per month
    number analyzed (Participants) | 75 | 77 | 152
    (all) | 1200 [500 to 2500] | 1500 [600 to 2500] | 1350 [590 to 2500]
Current BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Some participants did not wish to disclose this information.
  kg/m^2
    number analyzed (Participants) | 80 | 78 | 158
    (all) | 28.9 (4.2) | 28.9 (4.3) | 28.9 (4.3)
Pre-pregnancy BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: Some participants did not wish to disclose this information.
  kg/m^2
    number analyzed (Participants) | 80 | 77 | 157
    (all) | 26.1 (4.2) | 26.2 (4.1) | 26.2 (4.1)
Nightly sleep duration [Mean (Standard Deviation); unit: Hours] — Population: One participant did not wish to disclose this information.
  Hours
    number analyzed (Participants) | 81 | 80 | 161
    (all) | 7.8 (1.3) | 8.2 (1.3) | 8.0 (1.3)
In the last week, sleep onset position [Count of Participants; unit: Participants]
  Left | 41 | 46 | 87
  Supine | 12 | 8 | 20
  Right | 33 | 29 | 62
  Prone | 2 | 0 | 2
In the last week, waking position [Count of Participants; unit: Participants]
  Left | 30 | 32 | 62
  Supine | 22 | 18 | 40
  Right | 26 | 31 | 57
  Prone | 4 | 2 | 6
When not pregnant, sleep onset positions [Count of Participants; unit: Participants]
  Left | 6 | 7 | 13
  Supine | 25 | 26 | 51
  Right | 10 | 9 | 19
  Prone | 42 | 39 | 81
When not pregnant, waking positions [Count of Participants; unit: Participants]
  Left | 12 | 10 | 22
  Supine | 25 | 29 | 54
  Right | 15 | 14 | 29
  Prone | 32 | 27 | 59
Part of bed sleeps on [Count of Participants; unit: Participants]
  Left | 42 | 31 | 73
  Right | 30 | 35 | 65
  Center | 11 | 12 | 23
Pillow use [Count of Participants; unit: Participants]
  None | 3 | 6 | 9
  Under head | 74 | 71 | 145
  Between knees | 7 | 5 | 12
  Under tummy | 4 | 0 | 4
  Behind back | 4 | 4 | 8
  Pregnancy pillow | 1 | 0 | 1
  Other (under feet or legs) | 2 | 6 | 8
Sleeps with bed partner [Count of Participants; unit: Participants] — Population: Some participants did not wish to disclose this information.
  Participants
    number analyzed (Participants) | 82 | 78 | 160
    (all) | 65 | 61 | 126
Uses insecticide treated bed net [Count of Participants; unit: Participants] — Population: Some participants did not wish to disclose this information.
  Participants
    number analyzed (Participants) | 81 | 78 | 159
    (all) | 19 | 17 | 36
Snores ≥3 nights per week [Count of Participants; unit: Participants] — Population: Some participants did not wish to disclose this information.
  Participants
    number analyzed (Participants) | 81 | 77 | 158
    (all) | 9 | 7 | 16
Past medical complications [Count of Participants; unit: Participants] | 4 | 2 | 6

OUTCOME MEASURES:

1. Primary Outcome: Birthweight of Baby
Description: Birthweight was measured using a Detecto newborn scale (Webb City, USA) and documented in the participant's hospital folder immediately after delivery by a midwife who was not a part of the study team and was not aware of the treatment allocation. Birthweight was subsequently abstracted by the blinded outcomes assessor.
  Analysis was by original assigned groups and on a complete-case basis (drop-outs excluded). The newborns included in the final analysis were born from November 31, 2015 through May 13, 2016.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: grams
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
grams | 3186 (484) | 3079 (493)

2. Primary Outcome: Birthweight Centile
Description: Birthweight centile was calculated using the Gestation-Related Optimal Weight (GROW) software,(1,2) which accounts for the main non-pathological factors affecting birthweight (gestational age, maternal height, maternal weight at booking, parity, ethnicity, and sex of the neonate) and, as such, enables delineation between constitutional and pathological smallness and more accurate detection of pregnancies at increased risk for adverse outcomes.(3,4) This was an additional trial outcome specified after trial commencement.
  1. Gardosi J, Francis A. Customized Weight Centile Calculator. Gestation Network; 2016. Available from: www.gestation.net
  2. Gardosi J, et al. Customised antenatal growth charts. Lancet. Elsevier; 1992 Feb;339(8788):283-7.
  3. Gardosi J. Horm Res. 2006;65(SUPPL. 3):15-8.
  4. Odibo A O, et al. J Matern Neonatal Med. 2011 Mar 10; 24(3):411-7.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: percent
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
percent | 43 [18 to 64] | 32 [14 to 60]

3. Secondary Outcome: Gestational Age at Delivery
Description: Gestational age at delivery (weeks) will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Median (Inter-Quartile Range); unit: Weeks
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Weeks | 39.1 [38.0 to 40.0] | 39.0 [38.1 to 40.3]

4. Secondary Outcome: Mode of Delivery
Description: Mode of delivery (unassisted, episiotomy, amniotomy, induced, fetal monitoring, forceps delivery, vacuum extraction, Cesarean section) will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants
  Spontaneous vaginal | 50 | 38
  Caesarean section | 32 | 40
  Vacuum extraction | 0 | 2

5. Secondary Outcome: Sex of Newborn (Male/Female)
Description: Sex of the newborn will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants
  Male | 50 | 39
  Female | 32 | 41

6. Secondary Outcome: Stillbirth
Description: If a stillbirth occurs, it will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants | 0 | 1

7. Secondary Outcome: Low Birthweight
Description: Low birthweight is defined as a birthweight ≤ 2500 grams at birth.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants | 7 | 6

8. Secondary Outcome: Small for Gestational Age
Description: Small for gestational age is defined as a Gestation-Related Optimal Weight (GROW) birthweight centile ≤ 10%.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants | 12 | 18

9. Secondary Outcome: Preterm Delivery
Description: Preterm delivery was defined as a gestational age (in weeks) at birth of less than 37 weeks, 0 days.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants | 5 | 8

10. Secondary Outcome: Received ≥ 1 Obstetrical Diagnosis During Labor/Delivery
Description: Any relevant diagnosis/diagnoses made during labor/delivery (e.g., gestational diabetes, gestational hypertension, meconium aspiration) will be recorded in the participant's health record as a part of routine obstetric care at the Korle Bu Teaching Hospital.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for baseline characteristics
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 82 | 80
Participants | 31 | 41

11. Other Pre Specified Outcome: Medical Staff Questionnaire - Session Time Requirement
Description: How long it took (in minutes), on average, to complete the Introduction and Instruction for PrenaBelt session.
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: Three, of four, maternity personnel conducting the device introduction sessions answered this question on the maternity personnel questionnaire.
Measure: Mean (Full Range); unit: minutes
Groups:
- Maternity Personnel: At completion of recruitment, the maternity personnel completing the device introduction sessions completed a questionnaire eliciting their training level, professional experience, and perspectives on session duration, delivery method, and challenges.
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 3
minutes | 10 [5 to 25]

12. Other Pre Specified Outcome: Medical Staff Questionnaire - Session Delivery
Description: How the medical staff person delivered the Introduction and Instruction for PrenaBelt session (e.g., one-on-one, in a group setting, or both) and the staff person's preference for delivery.
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: All four maternity personnel conducting the device introduction sessions completed this question on the maternity personnel questionnaire.
Measure: Count of Participants; unit: Participants
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
Participants
  One-on-one | 1
  Group | 0
  Both | 3

13. Other Pre Specified Outcome: Medical Staff Questionnaire - Session Difficulties
Description: Did the medical staff person or the participants encounter any difficulties during the Introduction and Instruction for PrenaBelt sessions (yes/no; if yes, describe)
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
Participants
  Yes | 1
  No | 3

14. Other Pre Specified Outcome: Medical Staff Questionnaire - Session Cultural Issues
Description: Were any cultural issues encountered during the Introduction and Instruction for PrenaBelt sessions (yes/no; if yes, describe).
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
Participants
  Yes | 0
  No | 4

15. Other Pre Specified Outcome: Medical Staff Questionnaire - Professional Training Level
Description: The professional training level (e.g., nursing, midwifery) of the medical staff person.
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: as for outcome 12
Measure: Count of Participants; unit: Participants
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
Participants
  Nurse with diploma in public health | 1
  Nurse with diploma in midwifery | 3

16. Other Pre Specified Outcome: Medical Staff Questionnaire - Professional Experience
Description: The professional experience (years working as a professional) of the medical staff person.
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: Four maternity personnel conducting the device introduction sessions completed this question on the maternity personnel questionnaire.
Measure: Mean (Full Range); unit: years
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
years | 8.33 [4 to 29]

17. Other Pre Specified Outcome: Medical Staff Questionnaire - Professional Difficulty Rating
Description: In comparison to the medical staff person's training and experience, the difficulty rating of delivering the sessions on a scale from 1 to 10:
  1 = Easy - medical staff person could have completed the sessions without training and experience.
  5 = Medium difficulty - medical staff person needed to use some professional training and experience.
  10 = Very difficult - professional training and experience did not help medical staff person at all
Time Frame: From first Introduction and Instruction for PrenaBelt session until the last session (approximately 7 months)
Population: as for outcome 16
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Maternity Personnel
Number analyzed (Participants) | 4
units on a scale | 4 [1 to 5]

18. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Understanding
Description: When the participant was introduced to and instructed how to use the PrenaBelt by the medical staff, how difficult was it to understand the PrenaBelt?
  Check box categories:
  Easy - participant did not have to ask any questions. Medium - participant had some questions. Difficult - participant had many questions and could not understand it.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: Per protocol, the PrenaBelt User Feedback Questionnaire was only administered to participants in the Arms/Groups with the PrenaBelt (n=82). 55 of these 82 completed the Questionnaire. The BPS was not expected to affect responses to the Questionnaire, so these Arms/Groups with the PrenaBelt were combined. No arms are missing from the entered data.
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Easy | 51
  Medium | 1
  Difficult | 0
  No response | 3

19. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Learning
Description: When the participant was introduced to and instructed how to use the PrenaBelt by the medical staff, how difficult was it to learn how to use the PrenaBelt?
  Check box categories:
  Easy - participant did not have to ask any questions. Medium - participant had some questions. Difficult - participant had many questions and could not put the PrenaBelt on correctly.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Easy | 51
  Medium | 1
  Difficult | 0
  No response | 3

20. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - General Adherence Pattern
Description: Did the participant use the PrenaBelt regularly (almost every night)?
  Check box categories:
  Regularly throughout her entire third trimester. More regularly at the beginning and less at the end. Less regularly at the beginning and more at the end. Not regularly at any time.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Regularly throughout her entire third trimester | 11
  More regularly at the beginning, less at the end | 32
  Less regularly at the beginning, more at the end | 3
  Not regularly at any time | 5
  No response | 4

21. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Nights of Use Per Week
Description: When the participant was using the PrenaBelt, did she use it:
  Check box categories:
  Every night of the week. 6 nights per week. 7 nights per week. 5 nights per week. 4 nights per week. 3 nights per week. 2 nights per week.
  1 nights per week. Did not use it at all.
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Every night of the week. | 10
  6 nights per week. | 1
  5 nights per week. | 25
  4 nights per week. | 5
  3 nights per week. | 7
  2 nights per week. | 2
  1 nights per week. | 1
  Did not use at all. | 0
  No response. | 4

22. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Deterrents to Use
Description: Did anyone tell the participant to stop using the PrenaBelt or that she should not be using the PrenaBelt (yes/no; if yes, explain)
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Yes | 3
  No | 52

23. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Other Uses
Description: Did the participant or anyone else use the PrenaBelt for anything else during daily activities besides sleep (yes/no; if yes, explain).
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Yes | 0
  No | 55

24. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Perception of Effect on Sleep Position
Description: How does the participant think the PrenaBelt affected her sleep position.
  Check box categories:
  Participant didn't notice any difference in her sleep position Participant changed position more often. Participant spent more time sleeping on her left side. Participant woke up more often during the night when she was on her back, would roll back onto her left side, and fall asleep.
  Over time, participant learned to not sleep on her back and woke up less at night.
  In the mornings, participant always woke up on her left side.
  Other, please specify:
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Didn't notice a difference | 2
  Changed position more often | 15
  Spent more time sleeping on left | 26
  Woke up on back, turned to left, fell asleep | 21
  Learned not to sleep on back, woke up less often | 22
  In morning, always woke up on her left | 17
  Other | 0

25. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Perception of Effect on Sleep
Description: In general, did the participant notice anything else that was different about her sleep when using the PrenaBelt.
  Check box categories:
  Participant's sleep quality improved. Participant's sleep quality worsened. Participant's sleep duration became longer. Participant's sleep duration became shorter. During the day, participant felt more alert. During the day, participant felt more drowsy. Participant stopped snoring. Participant started snoring. Participant woke up less often throughout the night.
  Other, please specify:
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Count of Participants; unit: Participants
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
Participants
  Sleep quality improved | 32
  Sleep quality worsened | 2
  Sleep duration became longer | 6
  Sleep duration became shorter | 21
  During the day, participant felt more alert | 8
  During the day, participant felt more drowsy | 1
  Stopped snoring | 2
  Started snoring | 0
  Woke up less often throughout the night | 11
  Other | 4

26. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Satisfaction
Description: On a scale of 1 to 10, participant's level of satisfaction with the PrenaBelt.
  Note:
  1 = extremely dissatisfied 5-6 = acceptable 10 = extremely satisfied
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
units on a scale | 8 [6 to 8.5]

27. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Comfort
Description: On a scale of 1 to 10, participant's level of comfort while wearing and sleeping with the PrenaBelt.
  Note:
  1 = extremely uncomfortable 5-6 = acceptable 10 = extremely comfortable
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
units on a scale | 8 [6 to 9]

28. Other Pre Specified Outcome: PrenaBelt User Feedback Questionnaire - Intention for Future Use
Description: On a scale of 1 to 10, participant's intention to use the PrenaBelt during a subsequent pregnancy if it was available to her.
  Note:
  1 = participant would never use it again 5-6 = participant would consider using it again 10 = participant would certainly use it again
Time Frame: At delivery of baby (on average, 38 - 40 weeks gestation)
Population: as for outcome 18
Measure: Median (Inter-Quartile Range); unit: units on a scale
Arm/Group | PrenaBelt
Number analyzed (Participants) | 55
units on a scale | 8 [7 to 9]

29. Other Pre Specified Outcome: Sleep Diary - PrenaBelt Adherence
Description: Participants in all study arms will be instructed to use the PrenaBelt/sham-PrenaBelt ("device") every night for the remainder of the pregnancy and will be given a simple Sleep Diary to track their nightly device use. The sleep diary will be returned to the study personnel by the participant after the delivery of her baby. By checking the box in her sleep diary for each night she uses the device (and, conversely, not checking the box for each night she does not use the device), adherence (the proportion of nights the device was used) to device use will be calculated.
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: 143 participants (68 treatments, 75 shams) completed and returned the sleep diary.Two arms: PrenaBelt (participants with and without BPS) and Control (participants with and without BPS). BPS was not expected to affect body position. We did not intend readers would interpret this as 4 different treatments. No arms are missing from the entered data.
Measure: Mean (Standard Deviation); unit: % (#nights used/#nights in trial)
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 68 | 75
% (#nights used/#nights in trial) | 52 (25) | 56 (26)

30. Other Pre Specified Outcome: Sleep Diary - Number of Nights in Trial
Description: as for outcome 29
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Number of nights in trial
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 68 | 75
Number of nights in trial | 80 (14) | 76 (16)

31. Other Pre Specified Outcome: Sleep Diary - Number of Nights Used Device
Description: as for outcome 29
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: as for outcome 29
Measure: Mean (Standard Deviation); unit: Number of nights used device
Arm/Group | PrenaBelt | Control
Number analyzed (Participants) | 68 | 75
Number of nights used device | 42 (21) | 43 (22)

32. Other Pre Specified Outcome: Body Position Sensor Participant Adherence
Description: Body Position Sensor (BPS) data (position - left, right, supine, prone - and time stamp) will be collected from participants in the "PrenaBelt with BPS" and "Control with BPS" Arms when she returns the BPS to study personnel after the delivery of her baby.
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: Of 32 participants (16 PrenaBelt, 16 sham) in the BPS cohort, 23 (14 PrenaBelt, 9 sham) had complete datasets for analysis.
Measure: Median (Inter-Quartile Range); unit: % of days
Arm/Group | PrenaBelt With Body Position Sensor | Control With Body Position Sensor (BPS)
Number analyzed (Participants) | 14 | 9
% of days | 19 [13 to 40] | 33 [19 to 45]

33. Other Pre Specified Outcome: Body Position Sensor Participant Time Used Per Night
Description: as for outcome 32
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: hours
Arm/Group | PrenaBelt With Body Position Sensor | Control With Body Position Sensor (BPS)
Number analyzed (Participants) | 14 | 9
hours | 5.3 [4.7 to 5.6] | 5.4 [4.2 to 6.0]

34. Other Pre Specified Outcome: Body Position Sensor Participant Sleep Time by Position
Description: as for outcome 32
Time Frame: Throughout third trimester (on average, from 28 through 40 weeks gestation)
Population: as for outcome 32
Measure: Median (Inter-Quartile Range); unit: % of total sleep time
Arm/Group | PrenaBelt With Body Position Sensor | Control With Body Position Sensor (BPS)
Number analyzed (Participants) | 14 | 9
% of total sleep time
  Percentage sleep time left | 27 [17 to 33] | 31 [30 to 36]
  Percentage sleep time right (%) | 35 [28 to 39] | 34 [28 to 37]
  Percentage sleep time supine (%) | 45 [33 to 49] | 37 [32 to 43]

ADVERSE EVENTS:
Time Frame: September 7 2015 through May 13 2016. Participants were in the trial throughout the third trimester of pregnancy (28-40 weeks gestation), which is approximately 12 weeks. They were recruited between 26-30 weeks gestation and followed through the remainder of pregnancy (fortnightly from 28 weeks gestation until 36 weeks and then weekly until delivery), labor, and delivery. The mean number of days in the trial was 75.7 (standard deviation 16.7; minimum=25 days, maximum=119 days).
Description: Two arms: PrenaBelt (participants with and without the BPS) and Control (participants with and without the BPS). BPS was not expected to affect body position. We did not inappropriately combine the BPS and non-BPS arms of the PrenaBelt Arm and the Control Arm to turn four arms into two arms, and no arms are missing from the entered data. This was done for the sake of clarity.
Arm/Group | PrenaBelt | Control
All-Cause Mortality (participants affected / at risk) | 0/100 | 0/100
Serious Adverse Events (participants affected / at risk) | 6/100 | 13/100
Other Adverse Events (participants affected / at risk) | 35/100 | 34/100
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrenaBelt (N=100) | Control (N=100)
Stillbirth (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — Death of the fetus at gestation ≥28 weeks or birthweight ≥1000 grams.
Placental abruption (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 2 (2)
Acute gastroenteritis (Gastrointestinal disorders) | 0 (0) | 1 (1)
Intrauterine growth restriction (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1) — Defined as fetal weight less than the 10th percentile for gestational age as determined through an ultrasound.
Preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Severe preeclampsia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Antepartum hemorrhage (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Chorioamnionitis (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Failure to progress (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 3 (3)
Imminent eclampsia (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 3 (3)
Persistent occiput posterior position (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Unfavourable cervix (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Neonatal Intensive Care Unit admission (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 2 (2)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | PrenaBelt (N=100) | Control (N=100)
Worsened sleep quality (Pregnancy, puerperium and perinatal conditions) | 2 (2) | 1 (1) — Participants who reported worsened sleep quality on the PrenaBelt User Feedback Questionnaire.
Shorter sleep duration (Pregnancy, puerperium and perinatal conditions) | 22 (22) | 8 (8) — Participants who reported shorter sleep duration on the PrenaBelt User Feedback Questionnaire.
Felt more drowsy during the day (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — Participants who reported feeling more drowsy during the day on the PrenaBelt User Feedback Questionnaire.
Felt too hot while wearing the device (Product Issues) | 2 (2) | 3 (3) — Participants who reported feeling too hot while wearing the device (PrenaBelt/sham) on the PrenaBelt User Feedback Questionnaire.
Felt too itchy while wearing the device (Product Issues) | 1 (1) | 2 (2) — Participants who reported feeling too itchy while wearing the device (PrenaBelt/sham) on the PrenaBelt User Feedback Questionnaire.
Macrosomia (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Breech presentation (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 2 (2)
Cephalopelvic disproportion (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 3 (3)
Cord presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Cord prolapse (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Face presentation (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Failed vacuum extraction (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Fetal distress (Pregnancy, puerperium and perinatal conditions) | 3 (3) | 6 (6)
Meconium stained grade 2 liquor (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Moderate oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Multiple uterine fibroids (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Placental abnormality (nonspecific) (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Postterm pregnancy (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Preterm labour (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 1 (1)
Prolonged premature ruptured of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Reduced fetal movement (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Severe oligohydramnios (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Term premature rupture of membranes (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1)
Unexplained vaginal bleeding (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0)
Gastroesophageal reflux exacerbation (Gastrointestinal disorders) | 0 (0) | 1 (1) — This participant discontinued participation in the trial because she her gastroesophageal reflux was exacerbated while using the device.
Placenta previa (Pregnancy, puerperium and perinatal conditions) | 0 (0) | 1 (1) — This participant was disqualified from participation in the trial by the PI after placenta previa was discovered on ultrasound two weeks after she entered the study.
Felt too hot while wearing the device (Product Issues) | 0 (0) | 1 (1) — This participant discontinued participation in the trial because she felt too hot while wearing the device.
Uterine contractions (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) — This participant discontinued participation in the trial because she felt uterine contractions while using the device.
Vomiting (Gastrointestinal disorders) | 1 (1) | 0 (0) — This participant discontinued participation in the trial because she started vomiting after she wore the device.

LIMITATIONS AND CAVEATS:
Did not include a non-intervention control group. Determination of adherence to device use was largely subjective, relying mostly on participants' self-reports. Low adherence rates. May be under-powered to detect a clinically meaningful difference.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No